CLINICAL TRIAL: NCT06975475
Title: SHR-A1811 and THPy in First or Second Line for HER2 Positive Advanced Breast Cancer Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UH-SHR-A1811 and THPy
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: breast caner; HER2 positive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): Trastuzumab，pyrotinib，Nab-Paclitaxel in first line;SHR-A1811 in second line
  Interventions: Drug: SHR-A1811,tratuzumab,pyrotinib,Nab-Paclitaxel
- ARM B (Active Comparator): SHR-A1811 in first line;Trastuzumab，pyrotinib，Nab-Paclitaxel in second line
  Interventions: Drug: SHR-A1811,tratuzumab,pyrotinib,Nab-Paclitaxel

INTERVENTIONS:
Drug: SHR-A1811,tratuzumab,pyrotinib,Nab-Paclitaxel — SHR-A1811:4.8mg/kg tratuzumab:Initial 8mg/kg followed by 6mg/kg pyrotinib:320mg Nab-Paclitaxel:100-150mg/m2

SUMMARY:
The aim of this project is to evaluate whether the sequence of Trastuzumab，pyrotinib and Nab-Paclitaxel in first line followed by SHR-A1811 in second line is superior to the sequence of SHR-A1811 in first line followed by Trastuzumab，pyrotinib and Nab-Paclitaxel in second line for HER2 positive breast cancer brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Females ≥18 yrs old
2. Pathologically confirmed HER2-positive advanced breast cancer;
3. Newly diagnosed brain metastes,At least one measurable intracranial lesion
4. Not received any systemic treatment for advanced stage
5. Radiotherapy was allowed in patients with an urgent need for control of intracranial symptoms
6. Adequate function of major organs
7. Willing to join in this study, able to provide written informed consent, good compliance and willing to cooperate with follow-up.

Exclusion Criteria:

1.Has leptomeningeal metastasis or cystic metastatic lesions confirmed by MRI or lumbar puncture; 2.Existence of third space fluid (e.g. massive ascites, pleural effusion, pericardial effusion) that is not well controlled by effective methods, e.g. drainage; 3.Has received whole brain radiotherapy, chemotherapy, surgery within 2 weeks before first dose of study therapy; 4.Has known clinically significant lung disease, that is, moderate-to-severe lung disease which severely affects respiratory function, including but not limited to: idiopathic pulmonary fibrosis, pneumonitis. Prior ≥ grade 3 interstitial lung disease is not allowed to enrolment; 5.Has received full-dose anticoagulants or thrombolytics within 10 days before enrolment, or non-steroid anti-inflammatory drugs with platelet inhibition 6.Previous treatment with trastuzumab deruxtecan (DS-8201a) or any other antibody drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase 1 inhibitor; 7.Participated in other drug clinical trials within 4 weeks before admission; 8.Other malignant tumors, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma, have been diagnosed in the past five years.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS2 | 2 years
  Progression-free survival after two lines of treatment (PFS2)

SECONDARY OUTCOMES:
overall survival(OS) | 4 years
  Date of randomization until date of death due to any cause
Intracranial CNS progression-free survival | 2 years
  Time from randomization to progression of intracranial lesions
Progression-free survival | 2 years
  Time from randomization to disease progression
adverse event | 2 years
  The proportion of patients with adverse reactions according to CTCAE5.0

IPD SHARING:
Plan to Share IPD: No